CLINICAL TRIAL: NCT00017251
Title: A Phase I Study Of Genasense, A Bcl-2 Antisense Oligonucleotide, Combined With Carboplatin And Etoposide In Patients With Small Cell Lung Cancer
Brief Title: Combination Chemotherapy Plus Oblimersen in Treating Patients With Previously Untreated Extensive-Stage Small Cell Lung Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2012-02387; 10992A; N01CM17102 (NIH); CDR0000068667 (Registry Identifier: PDQ (Physician Data Query))
Record Dates: First submitted 2001-06-06; First posted 2003-01-27 (Estimated); Last update posted 2013-01-24 (Estimated); Status verified 2013-01

CONDITIONS: Extensive Stage Small Cell Lung Cancer
MeSH Terms: interventions — oblimersen; Carboplatin; Etoposide

ARMS (1):
- Treatment (oblimersen sodium, carboplatin, etoposide) (Experimental): Patients receive G3139 IV continuously on days 1-8, carboplatin IV over 30 minutes on day 6, and etoposide IV over 1 hour on days 6-8. Treatment repeats every 3 weeks for up to 6 courses in the absence of unacceptable toxicity or disease progression.
  Interventions: Biological: oblimersen sodium; Drug: carboplatin; Drug: etoposide; Other: pharmacological study; Other: laboratory biomarker analysis

INTERVENTIONS:
Biological: oblimersen sodium — Given IV
  Other Names: augmerosen; G3139; G3139 bcl-2 antisense oligodeoxynucleotide; Genasense
Drug: carboplatin — Given IV
  Other Names: Carboplat; CBDCA; JM-8; Paraplat; Paraplatin
Drug: etoposide — Given IV
  Other Names: EPEG; VP-16; VP-16-213
Other: pharmacological study — Correlative studies
  Other Names: pharmacological studies
Other: laboratory biomarker analysis — Correlative studies

SUMMARY:
Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Oblimersen may make tumor cells more sensitive to chemotherapy drugs. Phase I trial to study the effectiveness of combination chemotherapy and oblimersen in treating patients who have extensive-stage small cell lung cancer

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Determine the maximum tolerated dose of oblimersen when combined with standard dose carboplatin and etoposide in patients with previously untreated extensive stage small cell lung cancer.

II. Determine the toxicity and feasibility of this regimen in these patients. III. Determine potential antitumor activity of this regimen as assessed by objective response in these patients.

OUTLINE: This is a multicenter, dose-escalation study of oblimersen (G3139).

Patients receive G3139 IV continuously on days 1-8, carboplatin IV over 30 minutes on day 6, and etoposide IV over 1 hour on days 6-8. Treatment repeats every 3 weeks for up to 6 courses in the absence of unacceptable toxicity or disease progression.

Cohorts of 3-6 patients receive escalating doses of G3139 until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that at which 2 of 3 or 2 of 6 patients experience dose-limiting toxicity.

PROJECTED ACCRUAL: Approximately 6-12 patients will be accrued for this study within 5 months.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed extensive stage small cell lungcancer
* No active CNS disease

  * CNS metastasis allowed provided patient completed 1 course of CNS radiotherapy
* Performance status - ECOG 0-2
* Performance status - Karnofsky 60-100%
* More than 2 months
* WBC at least 3,000/mm^3
* Absolute neutrophil count at least 1,500/mm^3
* Platelet count at least 100,000/mm^3
* Bilirubin normal
* AST and ALT no greater than 2.5 times upper limit of normal (ULN)
* PT and PTT no greater than 1.5 times ULN
* Creatinine normal
* Creatinine clearance at least 60 mL/min
* No symptomatic congestive heart failure
* No unstable angina pectoris
* No cardiac arrhythmia
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* No prior allergic reactions to compounds of similar chemical or biologic composition to study agents
* No other uncontrolled concurrent illness
* No ongoing or active infection
* No psychiatric illness or social situation that would preclude study compliance
* See Disease Characteristics
* At least 1 week since prior CNS radiotherapy and recovered
* No prior radiotherapy to more than 25% of skeleton
* No other prior anticancer therapy
* No other concurrent investigational agents
* No other concurrent anticancer therapy
* No concurrent anticoagulation therapy
* No concurrent combination antiretroviral therapy for HIV-positive patients

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2001-04; Primary Completion 2004-01 (Actual)

PRIMARY OUTCOMES:
Feasibility and toxicity of the regimen monitored using the Common Toxicity Criteria Version 2.0 | Up to 3 years
  Data will be summarized separately for each dose level, by severity, and type of toxicity.
Maximally tolerated dose of oblimersen sodium | 8 days

SECONDARY OUTCOMES:
Potential antitumor activity (responses to therapy) | Up to 3 years
  Will be analyzed using simple descriptive statistics only.
Whether concomitant carboplatin and etoposide administration alters oblimersen sodium steady state level | Day 6 and 8
  Will be analyzed using a paired t-test. If there are outliers or the distribution of changes in oblimersen sodium levels appears to be highly non-normal, the data will be analyzed using the Wilcoxon singed-rank test.

CONTACTS AND LOCATIONS:
Overall Officials: Charles Rudin, Principal Investigator — University of Chicago Comprehensive Cancer Center
Locations (1):
- University of Chicago Comprehensive Cancer Center, Chicago, Illinois, United States